CLINICAL TRIAL: NCT07043465
Title: Ambulant Monitoring to Detect Hemodynamic and Electrical Impact of Severe Tricuspid Valve Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S68180
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Tricuspid Regurgitation (TR)
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14 days ambulatory rhtyhm monitoring (Experimental): 14 days ambulatory rhtyhm monitoring to detect electrical instability
  Interventions: Diagnostic Test: 14 days ambulatory rhythm monitoring

INTERVENTIONS:
Diagnostic Test: 14 days ambulatory rhythm monitoring — 14 days ambulatory rhythm monitoring using Byteflies

SUMMARY:
This exploratory study aims to study the feasibility to detect early signs of disease progression in patients with severe TVR (grade ≥3/4) by monitoring electrical cardiac activity and correlating it with echocardiographic findings. The Byteflies monitoring device will be used for continuous 14-day outpatient ECG tracking. Transthoracic echocardiography will assess structural and pressure changes in the heart and liver. The goal is to improve early detection of right heart failure and hepatic congestion.

ELIGIBILITY:
Inclusion Criteria:

* Tricuspid valve regurgitation (TVR) grade ≥3/4 documented on Colour Doppler during routine transthoracic echocardiography
* Normal sinus rhythm
* Dutch speaking

Exclusion Criteria:

* History of cardiac surgery
* Abnormal rhythm at baseline visit
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Atrial electrical instability | 14 days
  Burden (expressed in % of total number of beats) of isolated atrial extrasystoles, runs of atrial tachycardie (less than 30 seconds), and sustained atrial arrhythmia (lasting 30 seconds or longer). These findings will be correlated with echocardopgrahic measurements to detect electrical markers associated with the severity of tricuspid valve regurgitation.
Ventricular electrical instability | 14 days
  Burden (expressed in % of total number of beats) of isolated ventricular extrasystoles, runs of ventricular tachycardie (less than 30 seconds), and sustained ventricular arrhythmia (lasting 30 seconds or longer). These findings will be correlated with echocardopgrahic measurements to detect electrical markers associated with the severity of tricuspid valve regurgitation.

SECONDARY OUTCOMES:
Bradycardia | 14 days
  Prevalence (%) of bradycardia events on 14 day rhythm monitoring defined as any occurence of ventricular rhythms <30 beats per minute or high-degree AV block. These findings will be correlated with echocardopgrahic measurements to detect electrical markers associated with the severity of tricuspid valve regurgitation.
Adverse events associated with rhythm monitoring | 14 days
  Prevalence (%) of any interruption in 14 days rhythm monitoring due to adverse events with the Byteflies monitoring patch (skin rash, allergic reactions,...)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No